CLINICAL TRIAL: NCT03375021
Title: A Randomized, Double-Blind, Tw0-Period Crossover Study to Assess the Efficacy and Safety of the Ampakine® Compound, CX717, Versus Placebo in Adults With Attention-Deficit Hyperactive Disorder
Brief Title: CX717 in the Treatment of Adult ADHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RespireRx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CX717-05-ADHD
Record Dates: First submitted 2017-12-07; First posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD, ampakine, Phase II clinical trial
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — CX717; Contraceptives, Oral

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-Blind, Two-Period Crossover Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 200 mg of drug product or placebo in matching size 0 capsules
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Sequence 1 PL (Experimental): Eligible subjects were randomized to Sequence 1 PL in which they received placebo (P) followed by crossover to CX717 200 mg low dose (L) of active treatment
  Interventions: Drug: CX717 200 mg; Drug: Placebo
- Sequence 2 PH (Experimental): Eligible subjects were randomized to Sequence 2 PH in which they received placebo (P) followed by crossover to CX717 800 mg High dose (H) of active treatment
  Interventions: Drug: CX717 800 mg; Drug: Placebo
- Sequence 3 LP (Experimental): Eligible subjects were randomized to Sequence 3 LP in which they received CX717 200 mg Low dose (L) of active treatment followed by crossover to placebo (P)
  Interventions: Drug: CX717 200 mg; Drug: Placebo
- Sequence 4 HP (Experimental): Eligible subjects were randomized to Sequence 2 PH in which they received CX717 800 mg High dose (H) of active treatment followed by crossover to placebo (P)
  Interventions: Drug: CX717 800 mg; Drug: Placebo

INTERVENTIONS:
Drug: CX717 200 mg — CX717 200 mg capsules BID
  Other Names: Low Dose
  Arms: Sequence 1 PL; Sequence 3 LP
Drug: CX717 800 mg — CX717 4 X 200 mg capsules BID
  Other Names: High Dose
  Arms: Sequence 2 PH; Sequence 4 HP
Drug: Placebo — Placebo 200 mg or 800 mg capsules BID

SUMMARY:
A Randomized, Double-Blind, Two-Period Crossover Study to Assess the Efficacy And Safety of the Ampakine® Compound, CX717, versus Placebo in Adults with Attention-Deficit Hyperactivity Disorder

DETAILED DESCRIPTION:
This study examined the clinical efficacy, tolerability and safety of CX717 in the treatment of adults with ADHD. The study was a double-blind, 2-period crossover study that compared 2 different doses of CX717 with placebo. Subjects were randomized to 1 of 4 different treatment sequences: placebo - low dose; low dose - placebo; placebo - high dose; or high dose - placebo. Each treatment period was 3 weeks with a 2-week washout between treatment periods. The doses chosen were 200 mg b.i.d. and 800 mg b.i.d.

ELIGIBILITY:
Inclusion Criteria:

1. Subject had ADHD as established by the Adult ADHD Clinical Diagnostic Scale (ACDS) Version 1.2
2. Patients must have at least moderately severe ADHD symptoms:

   * Subject had an ADHD-RS score of ≥22
   * Subject had a CGI-S score of ≥4
3. Subject was male
4. Subject was 18 - 50 years old, inclusive
5. Subject could read well enough to understand the informed consent form and other patient materials.

Exclusion Criteria:

1. Subject had a DSM-IV diagnosis of ADHD not otherwise specified
2. Subject had a current or lifetime history of bipolar disorder or any psychotic disorder as established by the Structured Clinical Interview for DSM-IV (SCID) (12)
3. Subject had a current history of major depression, substance abuse or dependence, generalized anxiety disorder, obsessive compulsive disorder, panic disorder, or posttraumatic stress disorder as established by SCID
4. Subject had a history of epilepsy, seizures, syncope, unexplained blackout spell(s), head trauma with loss of consciousness, or febrile seizures
5. Subject had a currently active medical condition (other than ADHD) that in the opinion of the Investigator could interfere with the ability of subject to participate in the study
6. Subject had a history of development delay in milestones
7. By history, the subject had an IQ less than 80
8. In the opinion of the Investigator, the subject had not derived significant therapeutic benefit from 2 or more appropriately dosed ADHD therapies
9. Subject was currently taking medication specifically for treatment of ADHD symptoms (e.g., stimulants, atomoxetine, tricyclic antidepressants, or bupropion).

   NOTE: subjects were off of stimulants for 2 weeks and off non-stimulant ADHD therapies for 4 weeks prior to the Period 1 Baseline Visit. Subject did not have evidence of a discontinuation or withdrawal reaction.
10. Subject was currently taking an anti-depressant prescription medication (e.g., paroxetine, sertraline, venlafaxine, etc.) or St. John's Wort
11. Subject was currently taking an anti-convulsant medication (e.g., phenytoin, carbamazepine, lamotrigine, valproic acid, etc.) or anti-psychotic medication
12. Subject had a clinically relevant abnormality on Screening evaluation including physical examination, vital signs, ECG, or laboratory tests
13. Subject was currently taking on a chronic basis any medication known to be primarily metabolized by a route other than the cytochrome P450 system
14. Subject was unwilling to refrain from taking medications that may have interfered with the assessment of cognitive function. Examples included benzodiazepines, sedating anti-histamines, zolpidem, and zaleplon. Herbal preparations with effects on the central nervous system (e.g., St. John's Wort, melatonin) were prohibited. These medications and herbal preparations were also prohibited throughout the study.
15. Subject was unwilling to refrain from taking more than 1 unit of alcohol within 24 hours of the clinic visits
16. Subject had a Body Mass Index (BMI) of less than 18 or greater than 35. No waivers were allowed.
17. Subject reported passive or active suicidal ideation or intent
18. Subject was concurrently participating in another clinical research study or investigational drug trial or had participated within the past 1 month
19. Subject was at high risk of non-compliance in the Investigator's opinion

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2005-07-19 (Actual); Primary Completion 2006-01-10 (Actual); Study Completion 2006-01-10 (Actual)

PRIMARY OUTCOMES:
ADHD-RS | 3 Weeks
  Attention-Deficit Hyperactivity Disorder Rating Scale (ADHD-RS) with Prompts The ADHD-RS is an 18-item scale that assesses the severity ADHD symptoms based on the symptom list in the DSM-IV. It is administered by a qualified health care professional.
  Each item is rated 0 - 3 (0=not present and 3=severe). Thus the scale has a range from 0 to 54.

SECONDARY OUTCOMES:
ADHD-RS subscales | 3 Weeks
  Attention Deficit Hyperactivity Disorder Rating Subscales: hyperactivity consisting of items 1-4, 8-10, 17-18, and inattentiveness consisting of items 5-7 and 11-16.
CGI-I | 3 Weeks
  Clinical Global Impression of Improvement
HAM-A | 3 Weeks
  Hamilton Rating Scale of Anxiety
HAM-D | 3 Weeks
  Hamilton Rating Scale of Depression
PSQI | 3 Weeks
  Pittsburgh Sleep Quality Index
ESS | 3 Weeks
  Eppworth Sleepiness Scale
ADHD-SRS | 3 Weeks
  Attention Deficit Hyperactivity Disorder Self Rating Scale
SCWT | 3 Weeks
  Stroop Color and Word Test
CTMT | 3 Weeks
  Comprehensive Trail Making Test
CPT | 3 Weeks
  Continuous Performance Task
FBDS | 3 Weeks
  Forward and Backward Digit Span

CONTACTS AND LOCATIONS:
Overall Officials: Len Adler, MD, Principal Investigator — NYU School of Medicine

IPD SHARING:
Plan to Share IPD: No